CLINICAL TRIAL: NCT06834698
Title: Topical Steroid Treatment for Meatal Stenosis: Clinical Outcomes and Uroflowmetry Assessment of Treatment Success
Brief Title: Steroid Treatment for Meatal Stenosis
Status: Completed | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/243
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Meatal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Topical steroid
  Interventions: Drug: Betamethasone Cream
- Meatotomy
  Interventions: Procedure: meatotomy

INTERVENTIONS:
Drug: Betamethasone Cream — Betamethasone 0.1% cream was administered to the external meatus twice per day for a duration of 21 days.
  Groups: Topical steroid
Procedure: meatotomy — In the event of steroid therapy failure, a meatotomy was performed under general anesthesia. The procedure involved squashing the ventral aspect of the pinpoint meatus for approximately 3-5 millimeters for 10 seconds and then incising it. The mucosal margins were sutured with absorbable sutures to avoid renarrowing.
  Urethral catheterization was not employed, and the procedure was performed on an outpatient basis. Patients were discharged following urination.
  Groups: Meatotomy

SUMMARY:
The goal of this observational study is to learn about the efficacy of topical steroid treatment for meatal stenosis.

The main question it aims to answer is:

Is steroid therapy effective for treatment of meatal stenosis? Participants already treated for meatal stenosis will be included.

ELIGIBILITY:
Inclusion Criteria:

* Presence of meatal stenosis

Exclusion Criteria:

* Presence of any anatomical problem or history of surgery

Max Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — This study is about external urethral meatal stenosis, which is seen in boys.
Study Population: The study included patients who were treated for meatal stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
The number of patients who showed significant clinical improvement over the course of the study | 2 months
  The resolution of symptoms such as straining, hesitancy, interrupted voiding, thin urine stream, and storage symptoms (e.g., urgency, frequency, urge incontinence) along with improved urination were considered indicators of treatment success. All patients underwent assessment through physical examination and observation of the urinary stream during micturition.

SECONDARY OUTCOMES:
The number of participants who exhibited treatment-related improvements in voiding curve pattern and maximal urine flow rate, as assessed by uroflowmetry, which measures the free flow of urine during micturition | 2 months
  Uroflowmetry is a diagnostic test that evaluates the flow of urine during micturition (urination), providing valuable insights into bladder function and obstruction.
  The voiding curve pattern refers to the shape and flow characteristics of the urine stream during urination. A normal voiding pattern typically presents a bell shape, reflecting a steady and consistent flow of urine without interruptions. However, in certain conditions, such as urinary tract obstruction or bladder dysfunction, the voiding curve may become irregular, showing reduced flow or intermittent pauses. A plateau-shaped voiding curve is typically observed in conditions like meatal stenosis. Improvement in the voiding curve pattern following treatment indicates that urine flow has become more consistent and efficient.
  Maximal urine flow rate (Qmax) is the highest rate at which urine is expelled during micturition. This measurement is important for assessing bladder function and identifying potential urinary flow iss

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Ilhan Varank Training and Research Hospital, Istanbul, Sancaktepe, Turkey (Türkiye)